CLINICAL TRIAL: NCT01649037
Title: A Randomised, Open Label Study to Compare the Efficacy of Nor Adrenaline and Terlipressin vs Step up Terlipressin Therapy in Hepatorenal Syndrome
Brief Title: To Compare the Efficacy of Nor Adrenaline and Terlipressin vs Step up Terlipressin Therapy in Hepatorenal Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-AKI-01
Record Dates: First submitted 2012-07-21; First posted 2012-07-25 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2013-12

CONDITIONS: Hepatorenal Syndrome
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Norepinephrine; Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nor adrenaline and terlipressin (Experimental)
  Interventions: Drug: nor adrenaline and terlipressin
- step up terlipressin (Active Comparator)
  Interventions: Drug: step up terlipressin therapy

INTERVENTIONS:
Drug: nor adrenaline and terlipressin — IV bolus terlipressin at the dose of 0.5 to 1 mg every 6 hours with the maximum daily cumulative dose of 4 mg/day.
  Continuous IV infusion of NA starting at 0.5 mg/h with doubling of dose after every 4 hours in case of no response.[ No response defined as MAP < 10, or 4 hr Urine output < 200 ml] with maximum dose upto 3 mg/h.
  Arms: nor adrenaline and terlipressin
Drug: step up terlipressin therapy — IV bolus terlipressin starting at 1.5 mg every 6 hours with increase in dose by 0.5 mg/6 hours in case of no response [< 25% decrease in s.creatinine] after every 48 hours. Maximum daily cumulative dose of 12 mg/day.
  Arms: step up terlipressin

SUMMARY:
All consecutive patients with liver cirrhosis having Acute Kidney Injury at admission or during hospitalization will be included in the study.

The diagnosis of liver cirrhosis will be based on the clinical grounds including Laboratory tests, endoscopic evidence, imaging (Ultrasonography/computed tomography) findings, and liver histology, when available.

ELIGIBILITY:
Inclusion Criteria:

- Patients with Liver cirrhosis and acute kidney injury. Patients consented for the study protocol by signing the informed consent.

Exclusion Criteria:

- Age less than 18 years Cirrhotics with kidney injury managed as outpatients. Patients undergoing renal replacement therapy (hemodialysis/renal transplantation).

Post liver transplantation patients. Hepatocellular carcinoma. History of coronary artery disease, ischaemic cardiomyopathy, ventricular arrhythmia, or peripheral vascular disease.

Patients with obstructive uropathy. Patient who withdrew or non complaint to the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the Response to treatment in each intervention group | 2 years

SECONDARY OUTCOMES:
Survival | 15 days
Side effects of the drug | 3 months
Complications and the predictors of the treatment response | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India